CLINICAL TRIAL: NCT05790980
Title: Assessment of Quality of Life in Thalassemic Patients at Assiut University Hospital: A Single-center Experience
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Reham Abdelraheem, Assiut University, Assiut University
Other Study IDs: quality of life in thalassemia
Record Dates: First submitted 2023-02-15; First posted 2023-03-30 (Actual); Last update posted 2023-03-30 (Actual); Status verified 2023-03

CONDITIONS: Thalassemia
MeSH Terms: conditions — Thalassemia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective

INTERVENTIONS:
Device: Abdominal ultrasound — Abdominal US to exclude splenomegaly and hepatomegaly or liver cirrhosis Echocardiology to show cardiac dysfunction
  Other Names: Echocardiology

SUMMARY:
The thalassemias are a group of inherited hematologic disorders caused by defects in the synthesis of one or more of the hemoglobin chains [1]. Thalassemia are classified into the alpha (α) and (β) thalassemia, which contain deficits in (α) and (β) globin production respectively (α)thalassemia are caused by decreased production of alpha-globin chains from chromosome 16. There are 4 types of (α) thalassemia: thalassemia silent carrier thalassemia carrier . Hemoglobin H disease thalassemia major Beta-thalassemia are caused by point mutations or more rarely deletions in the β-globin gene on chromosome 11, leading to reduced (β+) or absent (β0) synthesis of the β chains of hemoglobin. Imbalances of globin chains cause hemolysis and impair erythropoiesis [4-7]. β-thalassemia can be classified into: Beta Thalassemia major, Beta Thalassemia intermedia, Beta Thalassemia minor Thalassemia is a chronic disease that presents a range of serious clinical and psychological challenges.

The effects of thalassemia on physical health can lead to physical deformity, growth retardation, and delayed puberty [9, 10]. Its impact on physical appearance, e.g., bone deformities and short stature, also contributes to a poor self-image [10, 11]. Severe complications such as heart failure, cardiac arrhythmia, liver disease, endocrine complications, and infections are common among thalassemia patients [8, 12].

DETAILED DESCRIPTION:
The problems mentioned do not only affect patients' physical functioning but also their emotional functioning, social functioning and school functioning, leading to impaired Health-related quality of life (HRQOL) of the patients [13]. QOL is a phrase used to refer to an individual's total wellbeing. This includes all emotional, social, and physical aspects of the individual's life. Health-related quality of life (HRQOL) Moreover, the term health-related quality of life (HRQOL) is often described as: "A term referring to the health aspects of quality of life, generally considered to reflect the impact of disease and treatment on disability and daily functioning; it has also been considered to reflect the impact of perceived health on an individual's ability to live a fulfilling life.[18-19] HRQOL is comprised of a number of dimensions of influence. Seven are commonly agreed upon

1. Physical well-being: the experience of physical symptoms such as pain, dyspnea, or nausea.
2. Functional well-being: the ability to participate in normal daily activities such as work and leisure pursuits.
3. Emotional well-being: this is comprised of both positive affective states (e.g. happiness, peace of mind) and negative affective states (e.g. sadness, anxiety).
4. Family well-being: the ability to maintain family relationships and communication.
5. Social functioning: the ability to participate and enjoy social roles and activities.[20]
6. Treatment satisfaction: including financial concerns.
7. Sexuality/intimacy: including concerns about body image.

ELIGIBILITY:
Inclusion Criteria:

* Thalassemic patients more than 18 years old.

Exclusion Criteria:

* Thalassemic patients less than 18 years old. Patients with other causes of aneamia. Patients with other causes of liver cirrhosis. Patients with other causes of renal diseases.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Thalassemic patients more than 18 years old.
Sampling Method: Non-Probability Sample
Enrollment: 68 (Estimated)
Dates: Start 2023-04-01 (Estimated); Primary Completion 2025-03-01 (Estimated); Study Completion 2025-06-01 (Estimated)

PRIMARY OUTCOMES:
Assisment of Quality of life in thalassemic patient | baseline
  assess the health-related quality of life among thalassemic patients attending Clinical hematology unit, Assiut University Hospital in a questionnaire manner

REFERENCES:
- [Background] Khodashenas M, Mardi P, Taherzadeh-Ghahfarokhi N, Tavakoli-Far B, Jamee M, Ghodrati N. Quality of Life and Related Paraclinical Factors in Iranian Patients with Transfusion-Dependent Thalassemia. J Environ Public Health. 2021 Aug 18;2021:2849163. doi: 10.1155/2021/2849163. eCollection 2021. PMID 34457009
- [Background] Shafique F, Ali S, Almansouri T, Van Eeden F, Shafi N, Khalid M, Khawaja S, Andleeb S, Hassan MU. Thalassemia, a human blood disorder. Braz J Biol. 2021 Sep 3;83:e246062. doi: 10.1590/1519-6984.246062. eCollection 2021. PMID 34495151
- [Background] Galanello R, Cao A. Gene test review. Alpha-thalassemia. Genet Med. 2011 Feb;13(2):83-8. doi: 10.1097/GIM.0b013e3181fcb468. No abstract available. PMID 21381239